CLINICAL TRIAL: NCT02670096
Title: A Single-center Pilot Study Evaluating the Immediate Effects of Low-dose Acetazolamide on Respiratory Control in Subjects With Treatment Emergent Sleep Disordered Breathing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00756
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Sleep Apnea
Keywords: acetazolamide; Treatment Emergent Sleep Disordered Breathing; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reference therapy (Experimental): * Baseline evaluation of subjects without acetazolamide administration
  * Follow up evaluation of subjects one hour after acetazolamide administration
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — Two single dose administrations of acetazolamide (once before daytime testing, and once before nighttime testing)
  Other Names: Diamox

SUMMARY:
This is a single center pilot study evaluating the immediate effects of low-dose acetazolamide on respiratory control in subjects with treatment emergent sleep disordered breathing. The purpose of this study is to assess the immediate effect one-time low-dose acetazolamide on sleep breathing in (Treatment Emergent Sleep Disordered Breathing) TE-CSA subjects compared to subjects' baseline evaluation without acetazolamide. Investigators will also try to determine the immediate effect of one-time low-dose acetazolamide on subjects' resting ventilation and ventilatory response slope compared to subjects' baseline evaluation without acetazolamide.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to 80 years
* TE-CSA
* Subjects are capable of giving informed consent

Exclusion Criteria:

* Hypersensitivity to acetazolamide or other sulfonamides
* Intake of carbonic anhydrase inhibitors within the last 72 hours
* Intake of medication that influences breathing, sleep, arousal or muscle physiology
* Cheyne-Stokes respiration
* Heart failure
* Renal failure
* Liver failure
* Chronic hypercapnea
* Hyponatremia
* Hypokalemia
* Pregnancy
* Breastfeeding mothers
* Active drug/alcohol dependence or abuse history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Severity of Obstructive Sleep Apnea before and after acetazolamide administration using Laboratory Nocturnal Polysomnography | 60 Days
Total lung capacity before and after acetazolamide administration | 60 Days

SECONDARY OUTCOMES:
Gas composition with and without acetazolamide using Resting Ventilation Study (RVS) | 20 Minutes
Measure of ventilatory response to carbon dioxide (CO2) without and with acetazolamide | 15 Minutes
Measurement of Arterial Blood Gas (ABG) | 60 Days
Measurement of Venous Blood (VB) Analysis | 60 Days

CONTACTS AND LOCATIONS:
Overall Officials: David Rapoport, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States